CLINICAL TRIAL: NCT00821301
Title: Phase 1b Single Arm, Open Label, Multi-Center Study of Fluphenazine HCl Monotherapy in Relapsed or Relapsed-and-Refractory Multiple Myeloma
Brief Title: Study of Fluphenazine in Relapsed or Relapsed-and-Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immune Control (Industry)
Responsible Party: Stephen Roth, Ph.D., Immune Control Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM-CL2
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Fluphenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fluphenazine HCl — Fluphenazine HCl will be administered intravenously. To quickly reach and maintain the target bone marrow concentration for 18 hours, the study drug will be administered using 3 bolus injections (0, 6, and 12 hours). Fluphenazine will be dose-escalated according to a modified Fibonacci scheme, terminating in 40% increments. Treatments will be administered on days 1 and 8 of every 21 day cycle.
  Other Names: Prolixin

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of fluphenazine in patients with advanced multiple myeloma. The study will also describe the efficacy of this drug.

DETAILED DESCRIPTION:
This is a multicenter, dose-escalating, Phase 1b trial in patients with relapsed or relapsed-and-refractory multiple myeloma. Patients will be dosed on Days 1 and 8 of each 21 day cycle.

This study will be conducted in two parts. In Part 1, the MTD determining portion of the study, patients will be enrolled in cohorts of 3 patients at each dose level. At least 3 patients will complete 21 days at each dose level and will be evaluated for safety and tolerability before additional patients are treated at higher doses. Doses will be increased following a modified Fibonacci scheme.

In Part 2, twelve additional patients will be enrolled at the MTD determined in Part 1 (or the dose for the highest dose cohort completed if the MTD has not been reached) to further evaluate the safety, tolerability, and preliminary efficacy of this dose regimen.

Serum fluphenazine pharmacokinetic studies will be performed during the first cycle of the therapy in all Part 1 and Part 2 consenting patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of multiple myeloma that is relapsed or relapsed-and-refractory after at least 2 or more prior lines of therapy. Patients must have achieved at least minor response (MR) to at least one prior line of therapy
* Progressive disease must have occurred either during or subsequent to the patient's last treatment for multiple myeloma prior to the current enrollment
* Measurable disease defined by serum M-protein ≥1 g/dL, or urine light chain ≥200 mg/24 hours, or abnormal serum FLC ratio with involved FLC > 10 mg/dL provided serum FLC ratio is abnormal
* Age >18 years
* Eastern Cooperative Oncology Group (performance status of ≤20
* Life expectancy ≥12 weeks
* Signed written informed consent per institutional and federal regulatory requirements
* Did not receive chemotherapy (including systemic steroids), immunotherapy (interferon), Imids (thalidomide/lenalidomide), proteasome inhibitors (bortezomib), or radiotherapy for at least 21 days prior to Day 1 of Cycle 1
* Did not receive any investigational treatment for at least 28 days prior to study entry
* Absolute granulocyte count of ≥1,000/μL, platelet count ≥50,000/μL, and hemoglobin ≥8.0 g/dL, with no transfusion within the preceding 7 days
* Adequate liver function defined by a bilirubin value ≤2 times the upper limit of normal (ULN), and transaminases (AST and ALT) values ≤2.5 times ULN
* Adequate renal function defined by a creatinine clearance of ≥30 mL/min
* Adequate cardiac function defined by a left ventricular ejection fraction (LVEF) ≥40%, QTc <450 msec, and no evidence of clinically significant dysrhythmias on ECG
* Patient must have substantially recovered from clinically significant toxicities from prior therapies for multiple myeloma
* Fertile men and women must agree to use a medically effective contraception method throughout the treatment period. Premenopausal women of reproductive capacity and women less than 24 months post menopause must have a negative serum pregnancy test documented prior to study entry

Exclusion Criteria:

* Patients who never achieved at least minor response (MR) to at least one prior line of therapy
* Clinical spinal cord compression syndromes (unless patient has undergone treatment, for example, surgery or radiation therapy, and neurological findings are ≤ Grade 1 and patient is off corticosteroids for spinal cord edema or on a stable regimen of < 10 mg/day prednisone equivalent
* Clinical signs of brain involvement or leptomeningeal disease
* Plasma cell leukemia (plasma cells > 2000/cubic mm)
* Women who are pregnant or breast feeding
* Other serious illness or medical condition(s) (see protocol)
* Hypersensitivity to fluphenazine or other phenothiazines
* Currently being treated with hematopoietic growth factors other than erythropoietin (EPO). Treatment with hematopoietic growth factors may be started during the study with development, or worsening, of cytopenia
* Concurrent use of anticholinergics
* Concurrent use of phenothiazine and atypical antipsychotics
* Concurrent use of anti-seizure drugs, with the exception of gabapentin for treatment of neuropathy
* Grade 2 or higher persisting prior treatment-related neuropathy
* Concurrent use of systemic steroids with the exception of chronically administered steroids equivalent to ≤ 10 mg/day prednisone if patient has been on this therapy for ≥1month
* History of seizures or extrapyramidal symptoms
* History of other malignancies within the past 3 years, other than adequately treated non-melanoma skin cancer, or in situ carcinoma of the cervix, unless the other malignancy is quiescent and medical monitor approval is obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Tolerability of fluphenazine. | 21 day treatment cycle(s)

SECONDARY OUTCOMES:
Changes in serum and urine M-protein or free light chain concentrations determined using protein electrophoresis. | 21 day treatment cycle(s)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Silver, M.D., FACP, Study Director
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Cancer Therapy and Research Center at the UT Health Sciences Center at San Antonio, San Antonio, Texas